CLINICAL TRIAL: NCT02892526
Title: Wound Vitality Markers in Forensic Pathology
Acronym: PLAIES VITALES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/CPRC/PLAIES VITALES/MART
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Wound
MeSH Terms: conditions — Wounds and Injuries | interventions — Abdominoplasty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Cutaneous tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vital wounds: from abdominoplasty of alive persons
  Interventions: Other: Abdominoplasty with exeresis of cutaneous tissue
- Post-mortem wounds: from autopsy of deceased persons
  Interventions: Other: Collection of cutaneous tissue

INTERVENTIONS:
Other: Abdominoplasty with exeresis of cutaneous tissue
  Groups: Vital wounds
Other: Collection of cutaneous tissue
  Groups: Post-mortem wounds

SUMMARY:
The purpose is to determine intrinsic properties of various immunohistochemical markers (FVIIIra, CD15, CD30, tryptase, TNFα, IL-1β, TGFα et TGFβ1) for diagnosis of vital wound, alone and in association (evaluation of sensibility with surgery wounds and evaluation of specificity with post-mortem wounds).

Secondary purposes are to measure the minimum time to obtain a positive labeling in vital wounds, and to evaluate inter-observer reproducibility of vitality diagnosis with different markers. Expression of microRNA miR 9, miR 21 et miR 198 will be also studied.

ELIGIBILITY:
Inclusion Criteria:

Alive persons:

- Abdominoplasty

Deceased persons:

- Medico-scientific autopsy for diagnosis

Exclusion Criteria:

Alive persons:

* Fragmented sample with non-visible banks
* Cutaneous pathology

Deceased persons:

* Persons under protection
* Medico-legal obstacle
* Cutaneous pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated in Plastic and Reconstructive Surgery and Maxillofacial Surgery departments at CHRU Nancy for therapeutic abdominoplasty.
  Deceased patients, whose medico-scientific autopsies are performed for diagnosis in Anatomy and Pathological Cytology or Legal Medicine departments.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Sensibility of markers for vitality diagnosis | baseline
Specificity of markers for vitality diagnosis | baseline

SECONDARY OUTCOMES:
Minimum time to obtain a labeling (between incision and devascularization) | baseline
Coefficient of inter-observer correlation of vitality diagnosis (for reproducibility analysis) | baseline
Expression level of miR 9 by qRT-PCR | baseline
Expression level of miR 21 by qRT-PCR | baseline
Expression level of miR 198 by qRT-PCR | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Laurent MARTRILLE, Principal Investigator — Service de Médecine Légale - CHRU de Nancy
Locations (1):
- CHRU Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No